CLINICAL TRIAL: NCT03040999
Title: A Randomized Phase III Study of Pembrolizumab Given Concomitantly With Chemoradiation and as Maintenance Therapy Versus Chemoradiation Alone in Subjects With Locally Advanced Head and Neck Squamous Cell Carcinoma (KEYNOTE-412)
Brief Title: Study of Pembrolizumab (MK-3475) or Placebo With Chemoradiation in Participants With Locally Advanced Head and Neck Squamous Cell Carcinoma (MK-3475-412/KEYNOTE-412)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-412; MK-3475-412 (Other: MSD); 173640 (Registry Identifier: JAPIC-CTI); KEYNOTE-412 (Other: MSD); 2016-003934-25 (EudraCT Number)
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Results first posted 2023-06-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and Neck Squamous Cell Carcinoma; Programmed Cell Death Receptor 1 (PD-1); Programmed Cell Death Receptor Ligand 1 (PD-L1); Programmed Cell Death Receptor Ligand 2 (PD-L2); PD1; PD-1; PDL1; PD-L1; PDL2
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cisplatin; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Cisplatin + CRT (Experimental): Participants receive a priming dose of pembrolizumab before initiation of CRT (either accelerated or standard fractionation radiotherapy regimen). During CRT, participants receive 2 doses of pembrolizumab and up to 3 cycles of Cisplatin (2 cycles during accelerated and 3 cycles during standard fractionation radiotherapy). Participants also receive up to an additional 14 cycles of pembrolizumab alone as maintenance therapy for a total of 17 cycles of pembrolizumab. If cisplatin and/or radiation therapy is discontinued, the participant may continue on treatment with pembrolizumab.
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Radiation: Accelerated Fractionation (AFX) Radiotherapy; Radiation: Standard Fractionation (SFX) Radiotherapy
- Placebo + Cisplatin + CRT (Placebo Comparator): Participants receive placebo before initiation of CRT (either accelerated or standard fractionation radiotherapy regimen). During CRT, participants receive 2 doses of placebo and up to 3 cycles of Cisplatin (2 cycles during accelerated and 3 cycles during standard fractionation radiotherapy). Participants also receive up to an additional 14 cycles of placebo alone for a total of 17 cycles of placebo. If cisplatin and/or radiation therapy is discontinued, the participant may continue on treatment with placebo.
  Interventions: Drug: Placebo; Drug: Cisplatin; Radiation: Accelerated Fractionation (AFX) Radiotherapy; Radiation: Standard Fractionation (SFX) Radiotherapy

INTERVENTIONS:
Biological: Pembrolizumab — Administered as an intravenous (IV) infusion every 3 weeks (Q3W)
  Other Names: KEYTRUDA®
  Arms: Pembrolizumab + Cisplatin + CRT
Drug: Placebo — Normal saline or dextrose solution administered as an IV infusion Q3W
  Arms: Placebo + Cisplatin + CRT
Drug: Cisplatin — 100 mg/m^2 administered as an IV infusion Q3W
  Other Names: Platinol®; Platinol®-AQ
Radiation: Accelerated Fractionation (AFX) Radiotherapy — 70 Gray (Gy) given in 35 fractions over 6 weeks
Radiation: Standard Fractionation (SFX) Radiotherapy — 70 Gy given in 35 fractions over 7 weeks

SUMMARY:
The purpose of this study is to determine the efficacy and safety of pembrolizumab given concomitantly with chemoradiation (CRT) and as maintenance therapy versus placebo plus CRT in participants with locally advanced head and neck squamous cell carcinoma (LA HNSCC). The primary hypothesis is that pembrolizumab in combination with CRT is superior to placebo in combination with CRT with respect to event-free survival (EFS).

ELIGIBILITY:
Inclusion Criteria:

* Has a pathologically proven new diagnosis of oropharyngeal p16 positive, oropharyngeal p16 negative, or larynx/hypopharynx/oral cavity (independent of p16) squamous cell carcinoma. Participants with oral cavity tumors need to have unresectable disease. Participants with multiple synchronous tumors are not eligible for the study.
* Has provided tissue for Programmed Cell Death Receptor Ligand 1 (PD-L1) biomarker analysis from a core or excisional biopsy. If an excisional or incisional biopsy has been performed, participants remain eligible for the study provided the residual disease meets the staging criteria required for the trial (e.g., excisional biopsy of a lymph node with residual T4 primary). Prior surgical debulking, including tonsillectomy, for the head and neck cancer under study is not allowed.
* Has evaluable tumor burden (measurable and/or non-measurable tumor lesions) assessed by computed tomography scan or magnetic resonance imaging, based on RECIST version 1.1
* Is eligible for definitive CRT and not considered for primary surgery based on investigator decision
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 performed within 10 days prior to receiving the first dose of study therapy
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study therapy
* Female and male participants of reproductive potential must agree to use adequate contraception throughout the study period and for up to 180 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating or has participated in a study with an investigational agent or using an investigational device within 4 weeks of the first dose of study therapy
* Has received prior therapy with an anti-Programmed Cell Death Receptor 1 (PD-1), anti-PD-L1, anti-Programmed Cell Death Receptor Ligand 2 (PD-L2) agent or with an agent directed to another co-inhibitory T-cell receptor or has previously participated in clinical studies with pembrolizumab
* Has received a live vaccine within 30 days prior to the first dose of study therapy
* Has cancer outside of the oropharynx, larynx, and hypopharynx or oral cavity, such as nasopharyngeal, sinus, other para-nasal, or other unknown primary head and neck cancer
* Has had prior systemic therapy, targeted therapy, radiotherapy treatment or radical surgery for head and neck cancer under study
* Has not recovered from major surgery prior to starting study therapy
* Has known active Hepatitis B or C
* Has known history of Human Immunodeficiency Virus (HIV)
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study therapy
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy is not considered a form of systemic treatment.
* Has history of a diagnosed and/or treated hematologic or primary solid tumor malignancy, unless in remission for at least 5 years prior to randomization
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has had previous allogeneic tissue/solid organ transplant
* Has active infection requiring systemic therapy
* Has a history of severe hypersensitivity reaction to pembrolizumab, Cisplatin or radiotherapy or their analogs
* Is pregnant or breast feeding or expecting to conceive or father children throughout the study period and for up to 180 days after the last dose of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2024-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (151):
- United States (24):
  - UCLA Medical Center ( Site 0273), Los Angeles, California
  - University of California San Francisco ( Site 0274), San Francisco, California
  - St. Joseph Heritage Healthcare ( Site 0254), Santa Rosa, California
  - Smilow Cancer Hospital at Yale New Haven ( Site 0256), New Haven, Connecticut
  - Rush University Medical Center ( Site 0260), Chicago, Illinois
  - Indiana University ( Site 0264), Indianapolis, Indiana
  - Mary Bird Perkins Cancer Center at St. Tammany Parish Hospital ( Site 0281), Baton Rouge, Louisiana
  - University of Massachusetts Memorial Medical Center ( Site 0285), Worcester, Massachusetts
  - University of Michigan Hospital and Health Systems ( Site 0267), Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute ( Site 0272), Detroit, Michigan
  - Mercy Clinic Cancer and Hematology - Chub O'Reilly Cancer Center ( Site 0290), Springfield, Missouri
  - St. Vincent Healthcare Frontier Cancer Center ( Site 0286), Billings, Montana
  - Comprehensive Cancer Centers of Nevada ( Site 8004), Las Vegas, Nevada
  - University of Rochester - James P. Wilmot Cancer Center ( Site 0255), Rochester, New York
  - Oncology Hematology Care, Inc. ( Site 8003), Cincinnati, Ohio
  - Willamette Valley Cancer Institute and Research Center ( Site 8000), Eugene, Oregon
  - St. Luke's Cancer Center - Anderson ( Site 0251), Easton, Pennsylvania
  - St. Francis Hospital Cancer Center ( Site 1461), Greenville, South Carolina
  - Texas Oncology-Arlington North ( Site 8005), Arlington, Texas
  - Texas Oncology-Austin Central ( Site 8002), Austin, Texas
  - Texas Oncology PA ( Site 8001), Longview, Texas
  - University of Virginia Health System ( Site 0261), Charlottesville, Virginia
  - Seattle Cancer Care Alliance/Univ of Washington Medical Center ( Site 0269), Seattle, Washington
  - Medical Oncology Associates (Summit Cancer Centers) ( Site 0257), Spokane, Washington
- Australia (6):
  - Blacktown Hospital Western Sydney Local Health District ( Site 0304), Blacktown, New South Wales
  - Liverpool Hospital ( Site 0301), Liverpool, New South Wales (Australia)
  - Princess Alexandra Hospital ( Site 0305), Brisbane, Queensland
  - Royal Brisbane and Women s Hospital ( Site 0302), Herston, Queensland
  - Royal Adelaide Hospital ( Site 0303), Adelaide, South Australia
  - Peter MacCallum Cancer Centre ( Site 0300), Melbourne, Victoria
- Austria (4):
  - Landeskrankenhaus - Universitatsklinikum Graz ( Site 0601), Graz
  - Krankenhaus der Barmherzigen Schwestern Linz ( Site 0603), Linz
  - Landeskrankenhaus Salzburg ( Site 0600), Salzburg
  - Allgemeines Krankenhaus der Stadt Wien ( Site 0602), Vienna/Wien
- Belgium (5):
  - Cliniques Universitaires Saint Luc - Bruxelles ( Site 0651), Brussels
  - UZ Gent ( Site 0650), Ghent
  - UZ Leuven Campus Gasthuisberg ( Site 0652), Leuven
  - C.H.U. Sart Tilman-Service d'Oncologie Medicale ( Site 0654), Liège
  - Clinique et Maternite Sainte-Elisabeth ( Site 0653), Namur
- Brazil (9):
  - Centro Regional Integrado de Oncologia ( Site 0002), Fortaleza, Ceará
  - Hospital Santa Izabel - Santa Casa de Misericordia da Bahia ( Site 0006), Salvador, Estado de Bahia
  - Liga Norte Riograndense Contra o Cancer ( Site 0005), Natal, Rio Grande do Norte
  - Hospital de Clinicas de Porto Alegre ( Site 0011), Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao ( Site 0001), Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos ( Site 0003), Barretos, São Paulo
  - Instituto do Cancer de Sao Paulo - ICESP ( Site 0004), São Paulo, São Paulo
  - Hospital das Clinicas da FMUSP de Ribeirao Preto ( Site 0008), Ribeirão Preto
  - Instituto Nacional do Cancer Jose Alencar Gomes da Silva INCA ( Site 0010), Rio de Janeiro
- Canada (8):
  - Tom Baker Cancer Centre ( Site 0063), Calgary, Alberta
  - Cross Cancer Institute ( Site 0064), Edmonton, Alberta
  - Juravinski Cancer Centre ( Site 0062), Hamilton, Ontario
  - London Health Sciences Centre ( Site 0055), London, Ontario
  - The Ottawa Hospital - Cancer Care ( Site 0052), Ottawa, Ontario
  - Princess Margaret Cancer Centre ( Site 0051), Toronto, Ontario
  - McGill University Health Centre ( Site 0061), Montreal, Quebec
  - CIUSSS de l Estrie - CHUS - Centre Hosp. Univ. Sherbrooke ( Site 0057), Sherbrooke, Quebec
- Colombia (4):
  - Hospital Pablo Tobon Uribe ( Site 0151), Medellín, Antioquia
  - Fundacion Valle del Lili ( Site 0150), Cali, Valle del Cauca Department
  - Centro Medico Imbanaco de Cali S.A ( Site 0156), Cali, Valle del Cauca Department
  - Centro de Investigacion Clinica del Country ( Site 0155), Bogotá
- Czechia (6):
  - FN Brno. ( Site 0703), Brno
  - Fakultni Nemocnice Hradec Kralove ( Site 0705), Hradec Králové
  - Fakultni nemocnice Olomouc ( Site 0701), Olomouc
  - Fakultni nemocnice Ostrava ( Site 0702), Ostrava
  - 2. LF UK a FN Motol ( Site 0704), Prague
  - Nemocnice Na Bulovce ( Site 0700), Prague
- France (5):
  - Centre Jean Bernard Laboratoire Mahe Meziani ( Site 0760), Le Mans
  - Clinique Francois Chenieux ( Site 0757), Limoges
  - Institut Claudius Regaud ( Site 0754), Toulouse
  - Institut De Cancerologie De Lorraine ( Site 0758), Vandœuvre-lès-Nancy
  - Institut Gustave Roussy ( Site 0759), Villejuif
- Germany (7):
  - Universitätsklinikum Erlangen ( Site 0801), Erlangen
  - SRH Waldklinikum Gera GmbH ( Site 0802), Gera
  - Universitares Cancer Center Hamburg - UCCH ( Site 0811), Hamburg
  - Medizinische Hochschule Hannover ( Site 0807), Hanover
  - Universitaetsklinikum Schleswig-Holstein-Campus Luebeck ( Site 0803), Lübeck
  - Klinikum der Universitaet Munchen ( Site 0810), München
  - Universitaetsklinik Ulm ( Site 0804), Ulm
- Israel (5):
  - Rambam MC ( Site 0903), Haifa
  - Hadassah Ein Karem Jerusalem ( Site 0902), Jerusalem
  - Rabin Medical Center ( Site 0904), Petah Tikva
  - Sheba MC ( Site 0901), Ramat Gan
  - Tel Aviv Sourasky Medical Center ( Site 0900), Tel Aviv
- Italy (8):
  - Azienda Ospedaliero Universitaria di Modena Policlinico ( Site 0954), Modena, MO
  - Azienda Ospedaliero Universitaria Careggi ( Site 0955), Florence
  - Istituto Nazionale Tumori ( Site 0950), Milan
  - Istituto Europeo di Oncologia ( Site 0953), Milan
  - Azienda Ospedaliera San Paolo ( Site 0952), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 0951), Napoli
  - Istituto Oncologico Veneto ( Site 0957), Padua
  - Fondazione IRCCS - Policlinico San Matteo ( Site 0960), Pavia
- Japan (10):
  - National Cancer Center Hospital East ( Site 0350), Kashiwa, Chiba
  - Hokkaido University Hospital ( Site 0351), Sapporo, Hokkaido
  - Hyogo Cancer Center ( Site 0354), Akashi, Hyōgo
  - Kagawa University Hospital ( Site 0359), Kita-gun, Kagawa-ken
  - Miyagi Cancer Center ( Site 0353), Natori-shi, Miyagi
  - Chiba Cancer Center ( Site 0358), Chiba
  - Hiroshima University Hospital ( Site 0352), Hiroshima
  - Osaka International Cancer Institute ( Site 0355), Osaka
  - Medical Hospital, Tokyo Medical And Dental University ( Site 0356), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 0357), Tokyo
- Netherlands (5):
  - Noordwest Ziekenhuisgroep NWZ ( Site 1350), Alkmaar
  - VU Medisch Centrum ( Site 1352), Amsterdam
  - UMCG ( Site 1351), Groningen
  - UMC St. Radboud ( Site 1356), Nijmegen
  - Erasmus University Medical Center ( Site 1354), Rotterdam
- Capital & Coast District Health Board - Wellington Hospital ( Site 0400), Wellington, Newtown, New Zealand
- Poland (8):
  - Dolnoslaskie Centrum Onkologii. ( Site 1001), Wroclaw, Lower Silesian Voivodeship
  - Mazowiecki Szpital Onkologiczny ( Site 1015), Wieliszew, Masovian Voivodeship
  - Beskidzkie Centrum Onkologii im. Jana Pawla II ( Site 1005), Bielsko-Biala
  - Szpital Morski im. PCK. Szpitale Pomorskie Sp. Z o.o ( Site 1007), Gdynia
  - Centrum Onkologii. Instytut im. Marii Sklodowskiej-Curie ( Site 1010), Gliwice
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie ( Site 1008), Krakow
  - Zachodniopomorskie Centrum Onkologii ( Site 1013), Szczecin
  - Centrum Onkologii-Instytut im. Marii Sklodowskiej-Curie ( Site 1000), Warsaw
- South Korea (5):
  - Seoul National University Bundang Hospital ( Site 0453), Seongnam-si, Gyeonggi-do
  - Chungbuk National University Hospital ( Site 0454), Cheongju-si, North Chungcheong
  - Chungnam National University Hospital ( Site 0455), Daejeon
  - Severance Hospital Yonsei University Health System ( Site 0452), Seoul
  - Samsung Medical Center ( Site 0450), Seoul
- Spain (7):
  - H.U. Vall de Hebron ( Site 1052), Barcelona
  - Hospital Duran i Reynals ( Site 1053), L'Hospitalet de Llobregat
  - Hospital Doce de Octubre ( Site 1054), Madrid
  - Hospital Universitario Ramon y Cajal ( Site 1055), Madrid
  - Hospital Clinico San Carlos ( Site 1051), Madrid
  - Hospital Universitario Virgen de la Victoria ( Site 1056), Málaga
  - Hospital Gral Universitario de Valencia ( Site 1050), Valencia
- Taiwan (7):
  - Chang Gung Medical Foundation - Kaohsiung ( Site 0501), Kaohsiung City
  - Taichung Veterans General Hospital ( Site 0506), Taichung
  - National Cheng Kung University Hospital ( Site 0503), Tainan
  - National Taiwan University Hospital ( Site 0500), Taipei
  - MacKay Memorial Hospital ( Site 0505), Taipei
  - Taipei Veterans General Hospital ( Site 0504), Taipei
  - Linkou Chang Gung Memorial Hospital ( Site 0502), Taoyuan District
- Turkey (Türkiye) (8):
  - Basken Adana Dr.Turgut Noyan Uygulama ve Arastirma Merkezi ( Site 1103), Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 1102), Ankara
  - Ankara Sehir Hastanesi ( Site 1108), Ankara
  - Istanbul Universitesi Istanbul Tip Fakultesi ( Site 1100), Istanbul
  - Medipol Universite Hastanesi ( Site 1104), Istanbul
  - Medical Park Izmir Hastanesi ( Site 1109), Izmir
  - Kocaeli Universitesi Tip Fakultesi ( Site 1106), Kocaeli
  - Inonu Universitesi Tip Fakultesi ( Site 1101), Malatya
- United Kingdom (9):
  - Norfolk & Norwich University Hospital NHS Foundation Trust ( Site 1206), Norwich, Norfolk
  - University Hospital of North Staffordshire ( Site 1202), Stoke-on-Trent, Staffordshire
  - Ipswich Hospital ( Site 1207), Ipswich, Suffolk
  - St Bartholomew s Hospital ( Site 1205), London
  - The Royal Marsden Foundation Trust ( Site 1200), London
  - Imperial Healthcare NHS Trust Charing Cross Hospital ( Site 1204), London
  - Lancashire Teaching Hospitals NHS Foundation Trust ( Site 1208), Preston
  - University Hospital Southampton NHS Foundation Trust ( Site 1203), Southampton
  - Royal Marsden NHS Foundation Trust ( Site 1201), Sutton

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Machiels JP, Tao Y, Licitra L, Burtness B, Tahara M, Rischin D, Alves G, Lima IPF, Hughes BGM, Pointreau Y, Aksoy S, Laban S, Greil R, Burian M, Hetnal M, Delord JP, Mesia R, Taberna M, Waldron JN, Simon C, Gregoire V, Harrington KJ, Swaby RF, Zhang Y, Gumuscu B, Bidadi B, Siu LL; KEYNOTE-412 Investigators. Pembrolizumab plus concurrent chemoradiotherapy versus placebo plus concurrent chemoradiotherapy in patients with locally advanced squamous cell carcinoma of the head and neck (KEYNOTE-412): a randomised, double-blind, phase 3 trial. Lancet Oncol. 2024 May;25(5):572-587. doi: 10.1016/S1470-2045(24)00100-1. Epub 2024 Mar 29. PMID 38561010
- [Derived] Machiels JP, Tao Y, Burtness B, Tahara M, Licitra L, Rischin D, Waldron J, Simon C, Gregoire V, Harrington K, Alves GV, Figueiredo Lima IP, Pointreau Y, M Hughes BG, Aksoy S, Hetnal M, Ge JY, Brown H, Cheng J, Bidadi B, Siu LL. Pembrolizumab given concomitantly with chemoradiation and as maintenance therapy for locally advanced head and neck squamous cell carcinoma: KEYNOTE-412. Future Oncol. 2020 Jun;16(18):1235-1243. doi: 10.2217/fon-2020-0184. Epub 2020 Jun 3. PMID 32490686
- See also: Merck Clinical Trial Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26854&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled who had locally advanced (LA) head and neck squamous cell carcinoma (HNSCC) and who were eligible for definitive chemoradiation therapy (CRT) and not considered for primary surgery based on investigator decision; had an Eastern Cooperative Oncology Group performance score of 0 or 1; had no distant metastases; and no active autoimmune disease or infection requiring systemic therapy.
Groups:
- Pembrolizumab + CRT + Pembrolizumab: On Cycle 1 Day 1 (each cycle is 21 days), participants received a priming dose of 200 mg Pembrolizumab followed by 100 mg/m^2 Cisplatin PLUS 70 Gray (Gy) Radiotherapy (accelerated (AFX) or standard fractionation radiotherapy (SFX)) on Day 8 of Cycles 1, 2 and Cycle 3 (SFX RT regimen only). During CRT, participants received 2 doses of pembrolizumab (Day 1 of Cycles 2 and 3) and up to 3 cycles of Cisplatin (2 cycles during AFX and 3 cycles during SFX RT). Participants also received up to an additional 14 cycles of pembrolizumab alone as maintenance therapy for a total of 17 cycles of pembrolizumab (approximately 1 year). If cisplatin and/or radiation therapy was discontinued, the participant may continue on treatment with pembrolizumab.
- Placebo + CRT + Placebo: On Cycle 1 Day 1 (each cycle is 21 days), participants received placebo followed by 100 mg/m^2 Cisplatin PLUS 70 Gray (Gy) Radiotherapy (accelerated (AFX) or standard fractionation radiotherapy (SFX)) on Day 8 of Cycles 1, 2 and Cycle 3 (SFX RT regimen only). During CRT, participants received 2 doses of placebo (Day 1 of Cycles 2 and 3) and up to 3 cycles of Cisplatin (2 cycles during AFX and 3 cycles during SFX RT). Participants also received up to an additional 14 cycles of placebo alone as maintenance therapy for a total of 17 cycles of placebo (approximately 1 year). If cisplatin and/or radiation therapy was discontinued, the participant may continue on treatment with placebo.
Period: Overall Study
Arm/Group | Pembrolizumab + CRT + Pembrolizumab | Placebo + CRT + Placebo
Started (Randomized) | 402 | 402
Treated | 398 | 398
Completed | 233 | 213
Not Completed | 169 | 189
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 12 | 13
Not completed — Death | 155 | 171
Not completed — Physician Decision | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + CRT + Pembrolizumab | Placebo + CRT + Placebo | Total
Number analyzed (Participants) | 402 | 402 | 804
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (9.0) | 58.6 (7.8) | 58.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 73 | 144
  Male | 331 | 329 | 660
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 59 | 106
  Not Hispanic or Latino | 324 | 312 | 636
  Unknown or Not Reported | 31 | 31 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 54 | 48 | 102
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 314 | 313 | 627
  More than one race | 19 | 28 | 47
  Unknown or Not Reported | 3 | 2 | 5
Human Papilloma Virus (HPV) Status [Count of Participants; unit: Participants] — Participants were assessed for HPV status using immunohistochemistry (IHC) analysis with CINtec® p16 histology assay. Positive p16 expression was defined as a strong and diffuse nuclear and cytoplasmic staining in 70% or more of the tumor cells.
  Participants
    Positive | 109 | 104 | 213
    Negative | 293 | 298 | 591
Disease stage at baseline [Count of Participants; unit: Participants] — Disease status at baseline was done using the American Joint Committee on Cancer (AJCC) Staging manual for head and neck cancers. AJCC7 for patients enrolled before Jan 1, 2018, and AJCC8 for those enrolled on or after Jan 1, 2018. Stages progress from best (II) to worst prognosis (IVb). Stage II: Large tumor size and/or limited local spread; Stage III: Large tumor size and/or limited local spread and/or spread to neck lymph nodes (NLNs); Stage IVa: Moderately advanced locally and/or spread to NLNs; Stage IVb: Very advanced locally and/or spread to NLNs with extranodal extension.
  Participants
    AJCC7 III | 8 | 11 | 19
    AJCC7 IVA | 61 | 58 | 119
    AJCC7 IVB | 12 | 14 | 26
    AJCC8 II | 0 | 1 | 1
    AJCC8 III | 132 | 125 | 257
    AJCC8 IVA | 146 | 152 | 298
    AJCC8 IVB | 43 | 41 | 84

OUTCOME MEASURES:

1. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. Participants without documented death at the time of analysis were censored at the date the participant was last known to be alive. The non-parametric Kaplan-Meier method was used to estimate the survival curve in each treatment group.
Time Frame: Up to approximately 62 months
Population: All randomized participants based on the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + CRT + Pembrolizumab | Placebo + CRT + Placebo
Number analyzed (Participants) | 402 | 402
Months | NA [NA to NA] — NA = median, upper limit, and lower limit were not reached due to insufficient number of participants with an event. | NA [NA to NA] — NA = median, upper limit, and lower limit were not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + CRT + Pembrolizumab vs Placebo + CRT + Placebo; Test type: Superiority; p = 0.1997, Log Rank; One-sided p-value based on log-rank test stratified by human papilloma virus (HPV) status and overall cancer stage; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.71 to 1.15] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by HPV status and overall cancer stage

2. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered study drug and which does not necessarily have to have a causal relationship with the study drug. An AE is any sign, symptom, disease, or worsening of preexisting condition temporally associated with study therapy and irrespective of causality to study therapy. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 88 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + CRT + Pembrolizumab | Placebo + CRT + Placebo
Number analyzed (Participants) | 398 | 398
Participants | 398 | 397

3. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered study drug and which does not necessarily have to have a causal relationship with the study drug. An AE is any sign, symptom, disease, or worsening of preexisting condition temporally associated with study therapy and irrespective of causality to study therapy. The number of participants who discontinued study drug due to an AE is presented.
Time Frame: Up to approximately 15 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + CRT + Pembrolizumab | Placebo + CRT + Placebo
Number analyzed (Participants) | 398 | 398
Participants | 163 | 132

4. Secondary Outcome: Change From Baseline in European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (Item 29) Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the quality of life (QoL) of cancer patients. For Global Health Status (GHS) (Item 29), participants are asked "How would you rate your overall health during the past week?" Individual items are scored on a 7-point (1=very poor to 7=excellent). Raw scores for each scale are standardized into a range of 0 to 100 by linear transformation, with a higher score indicating a better level of function and better overall GHS. A change from baseline of 10 points on the 100-point EORTC QLQ-C30 scale is considered as clinically relevant. Analysis based on a constrained longitudinal data analysis (cLDA) model with the patient reported outcomes (PRO) scores as the response variable with covariates for treatment, time, treatment by time interaction, and stratification factors of human papilloma virus (HPV) status and overall cancer stage.
Time Frame: Baseline and up to week 45
Population: Participants with at least one patient reported outcome (PRO) assessment available for this specific endpoint and who had received at least 1 dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab + CRT + Pembrolizumab | Placebo + CRT + Placebo
Number analyzed (Participants) | 393 | 392
Scores on a scale | 1.93 [-0.12 to 3.99] | 6.17 [4.10 to 8.23]
Statistical Analysis 1: Comparison: Pembrolizumab + CRT + Pembrolizumab vs Placebo + CRT + Placebo; Difference in Least Squares Mean; Test type: Other; p = 0.0015, cLDA; Difference in Least squares mean = -4.24, 95% CI 2-sided [-6.85 to -1.63] — Based on a cLDA model with the PRO scores as the response variable with covariates for treatment, time, treatment by time interaction, and stratification factors of HPV status and overall cancer stage

5. Secondary Outcome: Change From Baseline in European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire-Head and Neck Questionnaire (EORTC QLQ-H&N35) Swallowing Score
Description: EORTC QLQ Head and Neck Questionnaire (H&N35) measures QoL in head and neck cancer (HNC) patients. It consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the swallowing scale (Items 35-38) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating more problems. Change from baseline in swallowing was measured. A change from baseline of 10 points on the 100-point EORTC QLQ-H&N35 is considered as clinically relevant. Analysis based on a cLDA model with the PRO scores as the response variable with covariates for treatment, time, treatment by time interaction, and stratification factors of HPV status and overall cancer stage.
Time Frame: Baseline and up to Week 45
Population: Participants with at least one PRO assessment available for this specific endpoint and who had received at least 1 dose of study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab + CRT + Pembrolizumab | Placebo + CRT + Placebo
Number analyzed (Participants) | 393 | 391
Scores on a scale | -3.86 [-6.57 to -1.15] | -3.35 [-6.08 to -0.62]
Statistical Analysis 1: Comparison: Pembrolizumab + CRT + Pembrolizumab vs Placebo + CRT + Placebo; Difference in Least Squares Mean; Test type: Other; p = 0.7719, cLDA; Difference in Least squares mean = -0.51, 95% CI 2-sided [-3.98 to 2.96] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Change From Baseline in European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire-Head and Neck Questionnaire (EORTC QLQ-H&N35) Speech Score
Description: EORTC QLQ Head and Neck Questionnaire (H&N35) measures QoL in head and neck cancer (HNC) patients. It consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the speech scale (Items 30-32) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating more problems. Change from baseline in speech was measured. A change from baseline of 10 points on the 100-point EORTC QLQ-H&N35 is considered as clinically relevant. Analysis based on a cLDA model with the PRO scores as the response variable with covariates for treatment, time, treatment by time interaction, and stratification factors of HPV status and overall cancer stage.
Time Frame: Baseline and up to Week 45
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab + CRT + Pembrolizumab | Placebo + CRT + Placebo
Number analyzed (Participants) | 393 | 391
Scores on a scale | -6.22 [-8.89 to -3.54] | -4.93 [-7.62 to -2.23]
Statistical Analysis 1: Comparison: Pembrolizumab + CRT + Pembrolizumab vs Placebo + CRT + Placebo; Difference in Least Squares Mean; Test type: Other; p = 0.4500, cLDA; Difference in Least squares mean = -1.29, 95% CI 2-sided [-4.64 to 2.06] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Change From Baseline in European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire-Head and Neck Questionnaire (EORTC QLQ-H&N35) Pain Symptom Score
Description: EORTC QLQ Head and Neck Questionnaire (H&N35) measures QoL in head and Neck Cancer (HNC) patients. It consists of 7 multi-item scales (pain in the mouth, problems with swallowing, senses, speech, social eating, social contact, and sexuality). Participant responses to the pain scale (Items 31-34) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating more problems. Change from baseline in pain symptoms was measured. A change from baseline of 10 points on the 100-point EORTC QLQ-H&N35 is considered as clinically relevant. Analysis based on a cLDA model with the PRO scores as the response variable with covariates for treatment, time, treatment by time interaction, and stratification factors of HPV status and overall cancer stage.
Time Frame: Baseline and up to Week 45
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab + CRT + Pembrolizumab | Placebo + CRT + Placebo
Number analyzed (Participants) | 393 | 391
Scores on a scale | -10.55 [-12.87 to -8.22] | -11.84 [-14.18 to -9.50]
Statistical Analysis 1: Comparison: Pembrolizumab + CRT + Pembrolizumab vs Placebo + CRT + Placebo; Difference in Least Squares Mean; Test type: Other; p = 0.3524, cLDA; Difference in Least squares mean = 1.29, 95% CI 2-sided [-1.43 to 4.02] — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: Change From Baseline in European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Physical Functioning Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the quality of life (QoL) of cancer patients. Participant responded to 5 questions from the EORTC QLQ-C30 about their physical functioning scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores were standardized, so that scores range from 0 to 100, where a higher score indicates a better physical functioning. A change from baseline of 10 points on the 100-point scale is considered as clinically relevant. Analysis was based on a cLDA model with the PRO scores as the response variable with covariates for treatment, time, treatment by time interaction, and stratification factors of HPV status and overall cancer stage.
Time Frame: Baseline and up to Week 45
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab + CRT + Pembrolizumab | Placebo + CRT + Placebo
Number analyzed (Participants) | 393 | 392
Scores on a scale | -5.58 [-7.37 to -3.80] | -3.53 [-5.32 to -1.74]
Statistical Analysis 1: Comparison: Pembrolizumab + CRT + Pembrolizumab vs Placebo + CRT + Placebo; Difference in Least Squares Mean; Test type: Other; p = 0.0963, cLDA; Difference in Least squares mean = -2.05, 95% CI 2-sided [-4.47 to 0.37] — [estimate comment as in outcome 4, analysis 1]

9. Primary Outcome: Event-free Survival (EFS)
Description: EFS was defined as the time from date of randomization to the date of first record of any of the following events: death due to any cause; progression per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by blinded independent central review (BICR) or biopsy as indicated for locoregional progression or recurrence or distant metastasis. As well as the first record of the following types of surgery: salvage surgery for persistent or residual disease at the primary tumor site requiring surgical removal when invasive cancer is present on final pathology; neck dissection or surgery (performed for clinical or radiological disease progression per RECIST 1.1) ≤ 20 weeks from end of CRT when invasive cancer is present; or neck dissection or surgery >20 weeks from end of CRT when invasive cancer is present. The non-parametric Kaplan-Meier method was used to estimate the EFS curve in each treatment group.
Time Frame: Up to approximately 62 months
Population: All randomized participants based on the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + CRT + Pembrolizumab | Placebo + CRT + Placebo
Number analyzed (Participants) | 402 | 402
Months | NA [44.7 to NA] — NA = median and upper limit not reached due to insufficient number of participants with an event. | 46.6 [27.5 to NA] — NA = upper limit not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + CRT + Pembrolizumab vs Placebo + CRT + Placebo; Test type: Superiority; p = 0.0429, Log Rank — P-value crossing boundary of 0.0242 required for statistical significance; One-sided p-value based on log-rank test stratified by human papilloma virus (HPV) status and overall cancer stage; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.68 to 1.03] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to approximately 88 months
Description: The population analyzed for all-cause mortality consisted of all randomized participants. The population for AEs consisted of all randomized participants who received ≥1 dose of study drug. Per protocol disease progression of cancer was not considered an AE unless related to study drug. Therefore, the following AE preferred terms not related to the drug were excluded: Neoplasm progression, Malignant neoplasm progression and Disease progression.
Arm/Group | Pembrolizumab + CRT + Pembrolizumab | Placebo + CRT + Placebo
All-Cause Mortality (participants affected / at risk) | 156/402 | 178/402
Serious Adverse Events (participants affected / at risk) | 245/398 | 197/398
Other Adverse Events (participants affected / at risk) | 398/398 | 396/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + CRT + Pembrolizumab (N=398) | Placebo + CRT + Placebo (N=398)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 24 (26) | 7 (7)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Achlorhydria (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 11 (11) | 12 (13)
Enterocolitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 2 (3) | 5 (6)
Nausea (Gastrointestinal disorders) | 17 (19) | 7 (8)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 5 (5) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 12 (12) | 12 (13)
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 15 (17) | 10 (11)
Asthenia (General disorders) | 2 (2) | 3 (3)
Chest pain (General disorders) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 8 (8)
Face oedema (General disorders) | 1 (1) | 1 (1)
Facial pain (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 4 (4)
Fibrosis (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 4 (4) | 3 (3)
Impaired healing (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 3 (3)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 10 (10) | 9 (9)
Swelling (General disorders) | 0 (0) | 1 (1)
Vascular device occlusion (General disorders) | 0 (0) | 1 (1)
Vascular stent thrombosis (General disorders) | 0 (0) | 1 (1)
Cholangitis sclerosing (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis fulminant (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 2 (2) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 4 (5) | 3 (3)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Candida sepsis (Infections and infestations) | 1 (1) | 0 (0)
Catheter site abscess (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 6 (6) | 3 (3)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Genitourinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B reactivation (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Infected fistula (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Oral bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 43 (49) | 25 (33)
Pneumonia aspiration (Infections and infestations) | 12 (12) | 5 (6)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (2)
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1)
Sepsis (Infections and infestations) | 12 (12) | 7 (7)
Septic shock (Infections and infestations) | 3 (3) | 2 (2)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 2 (2)
Stoma site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 2 (2) | 2 (2)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Systemic infection (Infections and infestations) | 2 (2) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 2 (3)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Tracheostomy infection (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1)
Urosepsis (Infections and infestations) | 1 (2) | 0 (0)
Vascular access site infection (Infections and infestations) | 0 (0) | 2 (2)
Vascular device infection (Infections and infestations) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (4)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrostomy failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation associated pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation necrosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (4) | 2 (3)
C-reactive protein increased (Investigations) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (6) | 5 (5)
Platelet count decreased (Investigations) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 3 (3) | 2 (2)
White blood cell count decreased (Investigations) | 3 (3) | 7 (9)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 9 (10) | 5 (6)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (10) | 3 (3)
Hypophagia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Tumour inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 5 (5) | 2 (4)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 33 (41) | 30 (33)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 5 (5)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epiglottic oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngeal necrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5)
Oropharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (5)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pharyngeal necrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia lipoid (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + CRT + Pembrolizumab (N=398) | Placebo + CRT + Placebo (N=398)
Anaemia (Blood and lymphatic system disorders) | 229 (298) | 205 (287)
Ear pain (Ear and labyrinth disorders) | 28 (29) | 33 (35)
Hypoacusis (Ear and labyrinth disorders) | 80 (84) | 49 (51)
Tinnitus (Ear and labyrinth disorders) | 75 (83) | 88 (92)
Hyperthyroidism (Endocrine disorders) | 40 (43) | 33 (35)
Hypothyroidism (Endocrine disorders) | 100 (110) | 54 (58)
Abdominal pain upper (Gastrointestinal disorders) | 22 (23) | 13 (13)
Constipation (Gastrointestinal disorders) | 179 (218) | 174 (213)
Diarrhoea (Gastrointestinal disorders) | 88 (121) | 82 (106)
Dry mouth (Gastrointestinal disorders) | 191 (206) | 173 (194)
Dyspepsia (Gastrointestinal disorders) | 26 (34) | 25 (26)
Dysphagia (Gastrointestinal disorders) | 177 (190) | 165 (185)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 30 (31) | 19 (21)
Nausea (Gastrointestinal disorders) | 222 (324) | 232 (337)
Odynophagia (Gastrointestinal disorders) | 87 (96) | 89 (98)
Oral pain (Gastrointestinal disorders) | 28 (30) | 22 (23)
Saliva altered (Gastrointestinal disorders) | 22 (23) | 26 (26)
Stomatitis (Gastrointestinal disorders) | 249 (279) | 232 (259)
Vomiting (Gastrointestinal disorders) | 131 (204) | 116 (168)
Asthenia (General disorders) | 74 (93) | 73 (89)
Fatigue (General disorders) | 126 (150) | 118 (137)
Localised oedema (General disorders) | 26 (29) | 28 (29)
Oedema peripheral (General disorders) | 21 (26) | 18 (20)
Pyrexia (General disorders) | 64 (94) | 43 (55)
Nasopharyngitis (Infections and infestations) | 14 (15) | 20 (20)
Oral candidiasis (Infections and infestations) | 77 (85) | 60 (71)
Pneumonia (Infections and infestations) | 23 (25) | 21 (23)
Urinary tract infection (Infections and infestations) | 26 (35) | 17 (21)
Radiation skin injury (Injury, poisoning and procedural complications) | 254 (260) | 242 (244)
Alanine aminotransferase increased (Investigations) | 79 (100) | 60 (74)
Aspartate aminotransferase increased (Investigations) | 59 (78) | 41 (49)
Blood creatinine increased (Investigations) | 92 (128) | 87 (129)
Gamma-glutamyltransferase increased (Investigations) | 47 (61) | 36 (40)
Lymphocyte count decreased (Investigations) | 95 (143) | 109 (147)
Neutrophil count decreased (Investigations) | 166 (228) | 152 (240)
Platelet count decreased (Investigations) | 97 (150) | 83 (120)
Weight decreased (Investigations) | 179 (192) | 183 (201)
White blood cell count decreased (Investigations) | 127 (224) | 135 (236)
Decreased appetite (Metabolism and nutrition disorders) | 104 (115) | 115 (126)
Dehydration (Metabolism and nutrition disorders) | 44 (49) | 38 (48)
Hyperglycaemia (Metabolism and nutrition disorders) | 31 (44) | 35 (51)
Hyperkalaemia (Metabolism and nutrition disorders) | 27 (38) | 36 (52)
Hyperuricaemia (Metabolism and nutrition disorders) | 31 (41) | 33 (50)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 41 (51) | 33 (41)
Hypocalcaemia (Metabolism and nutrition disorders) | 38 (48) | 31 (42)
Hypokalaemia (Metabolism and nutrition disorders) | 100 (142) | 74 (108)
Hypomagnesaemia (Metabolism and nutrition disorders) | 110 (163) | 96 (144)
Hyponatraemia (Metabolism and nutrition disorders) | 79 (109) | 71 (109)
Hypophosphataemia (Metabolism and nutrition disorders) | 30 (33) | 19 (32)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (34) | 28 (34)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (26) | 14 (14)
Neck pain (Musculoskeletal and connective tissue disorders) | 35 (38) | 36 (38)
Trismus (Musculoskeletal and connective tissue disorders) | 12 (14) | 23 (25)
Dizziness (Nervous system disorders) | 30 (42) | 24 (28)
Dysgeusia (Nervous system disorders) | 132 (137) | 134 (139)
Headache (Nervous system disorders) | 39 (46) | 49 (54)
Peripheral sensory neuropathy (Nervous system disorders) | 34 (36) | 39 (42)
Anxiety (Psychiatric disorders) | 22 (24) | 14 (14)
Insomnia (Psychiatric disorders) | 57 (61) | 43 (50)
Acute kidney injury (Renal and urinary disorders) | 52 (74) | 39 (53)
Cough (Respiratory, thoracic and mediastinal disorders) | 65 (75) | 64 (71)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 49 (52) | 62 (69)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (24) | 20 (26)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 32 (40) | 25 (32)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 25 (25)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 91 (98) | 72 (79)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 51 (52) | 48 (48)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 39 (45) | 42 (50)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (15) | 22 (23)
Dry skin (Skin and subcutaneous tissue disorders) | 17 (18) | 21 (21)
Erythema (Skin and subcutaneous tissue disorders) | 27 (28) | 19 (21)
Pruritus (Skin and subcutaneous tissue disorders) | 52 (57) | 27 (34)
Rash (Skin and subcutaneous tissue disorders) | 59 (70) | 24 (26)
Hypertension (Vascular disorders) | 21 (26) | 33 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT03040999/Prot_SAP_001.pdf